CLINICAL TRIAL: NCT06659705
Title: Cutting Edge Imaging for Earlier Pancreatic Cancer Diagnosis: Evaluation of Positron Emission Tomography (PET) With the Fibroblast Activation Protein Inhibitor (FAPI)
Brief Title: Cutting Edge Imaging With PET-FAPI for Earlier Pancreatic Cancer Diagnosis (INDIGO-FAPI)
Acronym: INDIGO-FAPI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2023-02
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Fibroblast Activation Protein Inhibitor; Positron Emission Tomography; Pancreatic ductal adenocarcinoma; PDAC; FAPI
MeSH Terms: interventions — FAPI-46; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort involving repeated medical imaging with a new radiotracer (FAPI) (Experimental): All patients of this study must have been previously enrolled in the HoMING cohort (NCT 04363983, sponsor APHP).
  Interventions: Drug: 68Ga-FAPI-46 for PET / CT scan and 177Lu-EB-FAPI for therapy

INTERVENTIONS:
Drug: 68Ga-FAPI-46 for PET / CT scan and 177Lu-EB-FAPI for therapy — Gallium 68-labeled fibroblast activation protein inhibitor (FAPI) used as radiotracer during PET imaging.

SUMMARY:
Assessment of the relevance of a new medical imaging test, FAPI PET, which could detect progression or relapse earlier than other tests currently available. Ultimately, it could enable early forms of pancreatic cancer to be detected and used for screening.

In addition to the usual examinations prescribed, FAPI PET scans will be repeated at several points in the treatment process.

All study patients must first have been included in the Homing cohort (NCT 04363983, APHP promotion). Clinical characteristics, judgement criteria and results of biological or imaging examinations carried out as part of this cohort will be shared.

Patient follow-up and participation in the study ends when conventional imaging (CT and MRI) shows disease progression, relapse or death.

DETAILED DESCRIPTION:
Development of imaging biomarkers derived from FAPI PET among patients with a newly-diagnosed resectable or locally advanced PDAC, in order (i) to detect a metastatic disease at inclusion and (ii) to detect disease recurrence after surgical resection with a higher sensitivity than the standard evaluation.

Prospective cohort involving repeated medical imaging with a new radiotracer (FAPI). Patients meeting inclusion criteria will be stratified according to the disease staging: resectable, borderline or locally advanced PDAC.

At inclusion after confirmed non-metastatic PDAC diagnosis, all patients will have:

Baseline exams (V1) with 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT (within 1 month after inclusion in HoMING study) for all enrolled patients with resectable, borderline or locally advanced PDAC at inclusion.

Second pre-operative exams (V1b) with 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT exams only for patients who received neoadjuvant/induction treatment.

Post-operative/Follow-up exams (V2 to V5) with 68Ga-FAPI-46 PET/CT starting 2 months after surgery (with or without neoadjuvant/induction treatment) or following the neoadjuvant/induction treatment even if the patient is eventually not eligible for surgery (+/-1 month), and then every 3 months (+/-1 month).

All patients of this study must have been previously enrolled in the HoMING cohort (NCT 04363983, sponsor APHP). Endpoints and clinical characteristics, as well as results of other biological or imaging exams (MRI, spectral and conventional CT), will be shared with the HoMING cohort.

The follow-up ends as soon as conventional CT images show a disease progression/recurrence.

Investigators and patients will be blinded for the results of FAPI. Patients will be followed-up according to the care schedule with no modification of patient management. When disease progression/recurrence is diagnosed by conventional CT scan (gold standard), FAPI PET imaging at earlier time points (t -3 months, -6 months…) will be post-hoc reviewed to see whether small lesions could have been detected.

ELIGIBILITY:
Inclusion Criteria:

1. Recent (<1 month) diagnosis of non-metastatic PDAC (cyto/histologically proven, non-metastatic on CT-scan and MRI)
2. Patient already enrolled in the HoMING prospective cohort (Sponsor: AP-HP, NCT04363983)
3. Age > 18 years old
4. Affiliation to a social security scheme
5. Signed informed consent

Exclusion Criteria:

1. Protected adults (guardianship, curatorship or safeguarding justice)
2. Pregnant or breastfeeding woman
3. Women of childbearing potential not using one highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-08-04 (Estimated); Study Completion 2030-08-08 (Estimated)

PRIMARY OUTCOMES:
EFS: Event Free Survival | 12 months
  Time from diagnosis to disease progression, recurrence or death (EFS: Event Free Survival). Radiomic features from the initial FAPI evaluation will be analyzed using univariable and multivariable survival models to detect and quantify statistical associations between feature values and EFS. A multivariable model will be proposed and will serve as basis for the estimation of screening sensitivity.

SECONDARY OUTCOMES:
Adverse Event during 68Ga-FAPI-46 PET/CT exams | 12 months
  Description the safety profile of 68Ga-FAPI-46 PET/CT exams
Evaluation of the tumor burden 68Ga-FAPI-46 PET/CT versus 18F-FDG PET/CT | 12 months
  Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT (Comparison of the tumor burden using the total FAP expression tumor volume/TFTV and the total metabolic tumor volume/TMTV*, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie -site Saint-Cloud, Saint-Cloud, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).